CLINICAL TRIAL: NCT05016960
Title: Sleep-SMART for Veterans With MCI and Insomnia: A Pilot Study
Brief Title: SleepSMART for Veterans With MCI and Insomnia
Acronym: SleepSMART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: D3721-P
Record Dates: First submitted 2021-08-13; First posted 2021-08-23 (Actual); Results first posted 2025-04-23 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-12

CONDITIONS: Insomnia; Mild Cognitive Impairment
Keywords: Insomnia; Mild Cognitive Impairment; Veterans; Behavioral Sleep treatment; CBT for Insomnia; CogSMART; Feasibility; Acceptability
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: The investigators will develop and pilot test a modified CBT-I treatment that incorporates technology, user-centered design principles, and CogSMART strategies to improve sleep and rehabilitation outcomes for Veterans with co-occurring insomnia and MCI. The investigators will assess the feasibility and acceptability of Sleep-SMART (Sleep Symptom Management and Rehabilitation Therapy), which will seamlessly incorporate select CogSMART cognitive strategies within a standard 6-session 50-minute CBT-I treatment protocol. Sleep-SMART will focus on enhancing CBT-I by providing supportive cognitive strategies designed to boost treatment learning and adherence.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sleep-SMART (Experimental): Sleep-SMART intervention
  Interventions: Behavioral: Sleep-SMART

INTERVENTIONS:
Behavioral: Sleep-SMART — Sleep-SMART is a telehealth delivered treatment for insomnia that follows the standard 6 session 50-minute Cognitive Behavioral Therapy for Insomnia (CBT-I) format. Sleep-SMART delivers CBT-I treatment along with training in select cognitive strategies from CogSMART to enhance intervention learning and adherence.

SUMMARY:
Cognitive Behavioral Therapy for Insomnia (CBT-I) is the first-line treatment for chronic insomnia. However, cognitive impairments may limit progress in CBT-I for older Veterans with Mild Cognitive Impairment (MCI). This study will develop and pilot test Sleep-SMART (Sleep Symptom Management and Rehabilitation Therapy), an adapted CBT-I treatment that incorporates Cognitive Symptom Management and Rehabilitation Therapy (CogSMART) principles with a goal of improving sleep treatment and rehabilitation outcomes for Veterans with co-occurring MCI and insomnia. The innovation of this study centers on enhancing CBT-I by providing supportive cognitive strategies designed to improve treatment adherence, learning, and acceptability. The investigators anticipate that by improving sleep it can concurrently improve daily functioning, increase quality of life, prevent or reduce late-life disability, and mitigate long-term cognitive decline in this Veteran population.

DETAILED DESCRIPTION:
Mild cognitive impairment (MCI) is an important public health concern for aging Veterans due to the increased risk for progression to dementia and increased mortality. Insomnia is common in MCI (occurring in up to 60% of patients) and increases risk for dementia, disability, and poor quality of life. Rates of MCI and insomnia are higher among Veterans than civilians, thus aging Veterans with MCI and comorbid insomnia represent a particularly high-risk population. The gold standard treatment for insomnia, Cognitive Behavioral Therapy for Insomnia (CBT-I), is a multi-component behavioral intervention. However, cognitive impairments experienced by individuals with MCI may limit the rate of progress in CBT-I. The use of memory support strategies can improve patient recall of therapeutic information, enhance treatment adherence, and improve treatment outcomes. Cognitive Symptom Management and Rehabilitation Therapy (CogSMART) provides compensatory strategies to improve learning, memory, attention, and executive functioning. CogSMART has been shown to improve cognition, functional capacity, neurobehavioral symptoms, and quality of life in diverse Veteran populations with cognitive impairment. Incorporating supportive CogSMART cognitive strategies into CBT-I has the potential to improve treatment learning, adherence, and outcomes for this Veteran population. This RR&D SPiRE research project will assist us in developing and evaluating Sleep-SMART (Sleep Symptom Management and Rehabilitation Therapy), an innovative user-informed approach for treatment of insomnia in Veterans with MCI. Sleep-SMART is intended to provide the core components of CBT-I along with training in compensatory cognitive strategies from CogSMART to enhance intervention adherence and learning. Provision of this supportive cognitive training will assist Veterans with cognitive impairments in maintaining compliance with the CBT-I regimen, thereby leading to faster and more complete treatment benefits. The principle aims for the investigation include: 1) developing the Sleep-SMART intervention and treatment manual; 2) assessing the feasibility and acceptability of Sleep-SMART in Veterans with MCI and insomnia; and 3) exploring the effects of Sleep-SMART on rehabilitation outcomes, quality of life, sleep, and cognitive functioning.

ELIGIBILITY:
Inclusion Criteria:

* Veterans ages 60 or older who are competent to provide informed consent
* Chart diagnosis of MCI based on previously published criteria
* DSM-5 diagnosis of insomnia and an Insomnia Severity Index (ISI) score >7 at baseline
* Ability to understand, speak, and read English with acceptable visual and auditory acuity

Exclusion Criteria:

* Sleep disorders other than insomnia as determined by medical chart review and clinical interview
* History of a neurological disorder, dementia, or moderate to severe TBI
* Auditory, visual, or other impairments that would prevent ability to use video teleconferencing or participate in assessments
* Schizophrenia, psychotic disorder, bipolar disorder, and/or current substance use disorder
* Suicidality more than "low risk" as assessed by the Columbia Suicide Severity Rating Scale

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-01-04 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erin Almklov, PhD, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (1):
- VA San Diego Healthcare System, San Diego, CA, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Veterans aged 60 or older with MCI and insomnia were recruited from VA San Diego health clinics between 12/07/2021 and 12/31/2023.
Pre-assignment Details: Enrolled participants were excluded from the treatment phase (phase 2) if they did not meet study eligibility criteria at pre-treatment assessment.
Groups:
- Phase 1 - Sleep-SMART Development: Phase 1 involved conducting a focus group with Veterans from the target population to inform development of the Sleep-SMART intervention and manual.
- Phase 2 - Sleep-SMART Treatment: Phase 2 involved piloting the Sleep-SMART treatment that was developed in Phase 1. Sleep-SMART is a telehealth-based treatment for insomnia that follows the standard 6 session 50-minute CBT-I format and delivers CBT-I treatment along with training in select CogSMART cognitive strategies to enhance intervention learning and adherence.
Period: Overall Study
Arm/Group | Phase 1 - Sleep-SMART Development | Phase 2 - Sleep-SMART Treatment
Started | 5 | 25
Completed | 4 | 16
Not Completed | 1 | 9
Not completed — Withdrawal by Subject | 1 | 9

BASELINE CHARACTERISTICS:
Population: Baseline and outcome data was not collected from Phase 1 participants as they did not participate in the SleepSMART treatment. Phase 1 participants completed a one time focus group interview which was conducted to help guide the development of the SleepSMART treatment protocol.
Groups:
- Phase 2 - Sleep-SMART Treatment: Participants in Phase 2 received the Sleep-SMART treatment intervention and were administered baseline measures. Baseline and outcome measures were not collected as part of Phase 1.
Arm/Group | Phase 2 - Sleep-SMART Treatment
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants] — Population: Data was analyzed for treatment completers (n=16).
  Participants
    number analyzed (Participants) | 16
    <=18 years | 0
    Between 18 and 65 years | 4
    >=65 years | 12
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data was analyzed for treatment completers (n=16).
  Participants
    number analyzed (Participants) | 16
    Female | 3
    Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data was analyzed for treatment completers (n=16).
  Participants
    number analyzed (Participants) | 16
    Hispanic or Latino | 1
    Not Hispanic or Latino | 14
    Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data was analyzed for treatment completers (n=16).
  Participants
    number analyzed (Participants) | 16
    American Indian or Alaska Native | 0
    Asian | 1
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 3
    White | 12
    More than one race | 0
    Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25
Insomnia Severity Index [Mean (Standard Deviation); unit: units on a scale] — Scores range from 0-28 with higher scores indicating more severe insomnia. Population: Data was analyzed for treatment completers (n=16)
  units on a scale
    number analyzed (Participants) | 16
    (all) | 19.40 (4.95)

OUTCOME MEASURES:

1. Primary Outcome: Client Satisfaction Questionnaire (CSQ-8)
Description: Self-report scale to assess level of client satisfaction for the intervention. Scores range from 8-32, higher score indicates higher satisfaction. Mean scores were calculated at post-treatment. No statistical analyses were performed.
Time Frame: At post-treatment (approximately 8 weeks from study enrollment). Note: study consenting and pre-treatment assessment occurred in week 1, followed by the 6-session SleepSMART treatment in weeks 2-7 and the post-treatment assessment in week 8.
Population: Note: Data was analyzed for 14 participants as 2 of the 16 treatment completers from phase 2 did not complete the outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Phase 2 - Sleep-SMART Treatment: Sleep-SMART is a telehealth-based treatment for insomnia that follows the standard 6 session 50-minute CBT-I format and delivers CBT-I treatment along with training in select CogSMART cognitive strategies to enhance intervention learning and adherence.
Arm/Group | Phase 2 - Sleep-SMART Treatment
Number analyzed (Participants) | 14
score on a scale | 29.43 (2.95)

2. Primary Outcome: Telehealth Usability Questionnaire (TUQ)
Description: Scale to assess the usability of telehealth to deliver the intervention. In this questionnaire, 1 - strongly disagree, 2 - disagree, 3 - somewhat disagree, 4 - neither agree nor disagree, 5 - somewhat agree, 6 - agree, 7 - strongly agree To determine the usability of the telehealth system, calculate the total and determine the average of the responses to all statements. The higher the overall average, the higher the usability of the telehealth system.
Time Frame: as for outcome 1
Population: Note: Data was analyzed for 13 participants as 3 of the 16 treatment completers from phase 2 did not complete the outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase 2 - Sleep-SMART Treatment
Number analyzed (Participants) | 13
score on a scale | 5.92 (1.15)

3. Primary Outcome: Acceptability of Intervention Measure (AIM)
Description: Rating scale assessing intervention acceptability; scores range from 1-5 with higher scores indicating higher levels of acceptability. Ratings were collected at post-treatment. Mean scores were calculated. No statistical analyses were performed.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase 2 - Sleep-SMART Treatment
Number analyzed (Participants) | 14
score on a scale | 4.39 (0.59)

4. Primary Outcome: Intervention Appropriateness Measure (IAM)
Description: Rating scale assessing intervention appropriateness; scores range from 1-5 with higher scores indicating higher levels of appropriateness. Mean scores were calculated. No statistical analyses were performed.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase 2 - Sleep-SMART Treatment
Number analyzed (Participants) | 14
score on a scale | 4.41 (.66)

5. Other Pre Specified Outcome: WHO Disability Assessment Schedule 2.0 (WHODAS 2.0)
Description: Self-report scale assessing Subjective level of disability. Scores range from 0-100, where 0 = no disability; 100 = full disability.
Time Frame: At pre-treatment and post-treatment. Note: study consenting and pre-treatment assessment occurred in week 1, followed by the 6-session SleepSMART treatment in weeks 2-7 and the post-treatment assessment in week 8.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase 2 - Sleep-SMART Treatment
Number analyzed (Participants) | 14
score on a scale
  Post treatment | 63.79 (16.192)
  Pre treatment | 62.50 (17.105)
Statistical Analysis 1: Comparison: Phase 2 - Sleep-SMART Treatment; Test type: Other — one group paired samples t test to compare scores at pre vs. post treatment; p = .503, t-test, 2 sided

6. Other Pre Specified Outcome: Quality of Life in Neurological Disorders (Neuro-QOL) Cognition Scale
Description: Self-report scales assessing subjective cognitive complaints and subjective everyday functioning. Each response option is assigned a value (e.g., 1=Not at all). To find the total raw score, sum the values of the response to each question. A higher Neuro-QoL score represents more of the concept being measured - higher scores indicate worse functioning for the cognition scale.
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase 2 - Sleep-SMART Treatment
Number analyzed (Participants) | 14
score on a scale
  Pre treatment | 24.86 (8.047)
  Post treatment | 26.57 (5.734)
Statistical Analysis 1: Comparison: Phase 2 - Sleep-SMART Treatment; Test type: Non-Inferiority — one group paired samples t test; p = .230, t-test, 2 sided

7. Other Pre Specified Outcome: Everyday Cognition Scale (ECoG)
Description: Collateral measure of cognitive and everyday functioning. Is a 39 item questionnaire used to measure a patient's cognitive function and aid in the detection and diagnosis of dementia and other neurodegenerative diseases that are associated with aging. Each item is answered on a 1-4 point scale with a minimum total raw score of 39 and a maximum score of 156. Higher score are indicative of worse functioning.
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase 2 - Sleep-SMART Treatment
Number analyzed (Participants) | 14
score on a scale
  Post treatment | 83.71 (30.19)
  Pre Treatment | 89.86 (34.576)
Statistical Analysis 1: Comparison: Phase 2 - Sleep-SMART Treatment; Test type: Other — one group paired samples t test; p = .061, t-test, 2 sided

8. Other Pre Specified Outcome: Insomnia Severity Index (ISI)
Description: Self-report scale assessing perceived insomnia severity; scores range from 0-28 with higher scores indicating more severe insomnia.
Time Frame: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase 2 - Sleep-SMART Treatment
Number analyzed (Participants) | 16
score on a scale
  Pre-treatment | 19.40 (4.95)
  End of treatment | 8.87 (6.89)
Statistical Analysis 1: Comparison: Phase 2 - Sleep-SMART Treatment; Test type: Other — one group paired samples t test; p < .001, t-test, 2 sided

9. Other Pre Specified Outcome: Pittsburgh Sleep Quality Index (PSQI)
Description: The Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire that assesses sleep quality over a one-month time interval. The Global PSQI score ranges from 0 to 21 with higher scores indicating poorer sleep quality.
Time Frame: as for outcome 5
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase 2 - Sleep-SMART Treatment
Number analyzed (Participants) | 13
score on a scale
  Pre-treatment | 11.69 (5.10)
  Post-treatment | 8.85 (3.16)
Statistical Analysis 1: Comparison: Phase 2 - Sleep-SMART Treatment; Test type: Other — one group paired samples t test; p = .01, t-test, 2 sided

10. Other Pre Specified Outcome: Wechsler Adult Intelligence Scale-IV (WAIS-IV) Digit Span (Total Raw Score)
Description: Performance based measure of auditory attention; raw scores range from 0-48 with higher scores indicating better performance.
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase 2 - Sleep-SMART Treatment
Number analyzed (Participants) | 14
score on a scale
  Pre-treatment | 22.79 (6.841)
  Post-treatment | 22.21 (6.739)
Statistical Analysis 1: Comparison: Phase 2 - Sleep-SMART Treatment; Test type: Other — one group paired samples t test; p = .625, t-test, 2 sided

11. Other Pre Specified Outcome: Brief Visuospatial Memory Test-Revised (Total Recall Raw Score)
Description: Performance based measure of Visual design learning and memory. Scores are based on individual performance and range from 0-36 with higher scores indicating better performance/memory.
Time Frame: as for outcome 5
Population: Note: Data was analyzed for 9 participants as 7 of the 16 treatment completers from phase 2 did not complete the outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase 2 - Sleep-SMART Treatment
Number analyzed (Participants) | 9
score on a scale
  Pre-treatment | 14.33 (5.454)
  Post-treatment | 16.00 (5.074)
Statistical Analysis 1: Comparison: Phase 2 - Sleep-SMART Treatment; Test type: Other — one group paired samples t test; p = .134, t-test, 2 sided

12. Other Pre Specified Outcome: Delis-Kaplan Executive Function System (D-KEFS) Trail Making Test (Condition: Number-letter Switching) Raw Score
Description: Performance based measures of attention, processing speed, and executive function. Scores are based on the time (number of seconds) to complete the task for the trail making test and range from <3 seconds to 240 seconds. Raw scores are presented in seconds with lower scores indicating better performance.
Time Frame: as for outcome 5
Population: Note: Data was analyzed for 8 participants as 8 of the 16 treatment completers from phase 2 did not complete the outcome measure.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Phase 2 - Sleep-SMART Treatment
Number analyzed (Participants) | 8
seconds
  Pre-treatment | 146.63 (46.745)
  Post-treatment | 140.13 (54.038)
Statistical Analysis 1: Comparison: Phase 2 - Sleep-SMART Treatment; Test type: Other — one group paired samples t test; p = .515, t-test, 2 sided

13. Other Pre Specified Outcome: Delis-Kaplan Executive Function System (D-KEFS) Verbal Fluency Test (Category Switching)
Description: Performance based measures of executive function (i.e., category switching total raw score). The task requires participants to alternate between generating words from two different semantic categories. Scores are based on the number of correct words generated. Total raw scores range from 0 to >21, with higher scores indicating better performance.
Time Frame: as for outcome 5
Population: Note: Data was analyzed for 12 participants as 4 of the 16 treatment completers from phase 2 did not complete the outcome measure.
Measure: Mean (Standard Deviation); unit: words generated
Arm/Group | Phase 2 - Sleep-SMART Treatment
Number analyzed (Participants) | 12
words generated
  Pre-treatment | 12.25 (2.417)
  Post-treatment | 11.75 (1.712)
Statistical Analysis 1: Comparison: Phase 2 - Sleep-SMART Treatment; Test type: Other — one group paired samples t test; p = .410, t-test, 2 sided

14. Other Pre Specified Outcome: Hopkins Verbal Learning Test-Revised (Delayed Recall Raw Score)
Description: Performance based measure of verbal list learning and memory (i.e., delayed recall raw score). Scores range from 0 to 12 with higher scores indicating better performance.
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: words recalled
Arm/Group | Phase 2 - Sleep-SMART Treatment
Number analyzed (Participants) | 14
words recalled
  Pre-treatment | 6.93 (3.13)
  Post-treatment | 7.14 (2.69)
Statistical Analysis 1: Comparison: Phase 2 - Sleep-SMART Treatment; Test type: Other — one group paired samples t test; p = .706, t-test, 2 sided

15. Other Pre Specified Outcome: Brief Visuospatial Memory Test-Revised (Delayed Recall Raw Score)
Description: Performance based measure of Visual design learning and memory. Scores are based on individual performance and range from 0 to 12. Higher scores indicate better performance/memory.
Time Frame: as for outcome 5
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: correctly recalled elements
Arm/Group | Phase 2 - Sleep-SMART Treatment
Number analyzed (Participants) | 9
correctly recalled elements
  Pre-treatment | 5.44 (2.5)
  Post-treatment | 6.56 (2.3)
Statistical Analysis 1: Comparison: Phase 2 - Sleep-SMART Treatment; Test type: Other — one group paired samples t test; p = .062, t-test, 2 sided

16. Other Pre Specified Outcome: Hopkins Verbal Learning Test-Revised (Total Immediate Recall Raw Score)
Description: Performance based measure of verbal list learning and memory (i.e., immediate recall raw score). Scores range from 0 to 36 with higher scores indicating better performance.
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: words recalled
Arm/Group | Phase 2 - Sleep-SMART Treatment
Number analyzed (Participants) | 14
words recalled
  Pre-treatment | 22.00 (5.55)
  Post-treatment | 21.0 (2.37)
Statistical Analysis 1: Comparison: Phase 2 - Sleep-SMART Treatment; Test type: Other — one group paired samples t test; p = .390, t-test, 2 sided

17. Other Pre Specified Outcome: Delis-Kaplan Executive Function System (D-KEFS) Trail Making Test (Condition: Number Sequencing)
Description: Performance based measures of attention, processing speed, and executive function. Scores are based on the time (number of seconds) to complete the task for the trail making test. Raw scores are presented in seconds with lower scores indicating better performance.
Time Frame: as for outcome 5
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Phase 2 - Sleep-SMART Treatment
Number analyzed (Participants) | 9
seconds
  Pre-treatment | 53.11 (17.43)
  Post-treatment | 47.33 (25.96)
Statistical Analysis 1: Comparison: Phase 2 - Sleep-SMART Treatment; Test type: Other — one group paired samples t test; p = .38, t-test, 2 sided

18. Other Pre Specified Outcome: Delis-Kaplan Executive Function System (D-KEFS) Trail Making Test (Condition: Letter Sequencing)
Description: as for outcome 17
Time Frame: as for outcome 5
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Phase 2 - Sleep-SMART Treatment
Number analyzed (Participants) | 9
seconds
  Pre-treatment | 65.22 (32.82)
  Post-treatment | 46.44 (15.75)
Statistical Analysis 1: Comparison: Phase 2 - Sleep-SMART Treatment; Test type: Other — One group paired samples t test; p = .064, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Deaths, serious adverse events, and non-serious adverse events were not assessed for this study.
Groups:
- Sleep-SMART: Sleep-SMART intervention
  Sleep-SMART: Sleep-SMART is a telehealth delivered treatment for insomnia that follows the standard 6 session 50-minute Cognitive Behavioral Therapy for Insomnia (CBT-I) format. Sleep-SMART delivers CBT-I treatment components along with training in select cognitive strategies from CogSMART to enhance intervention learning and adherence.
Arm/Group | Sleep-SMART
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-07-21): https://cdn.clinicaltrials.gov/large-docs/60/NCT05016960/Prot_001.pdf
  • Statistical Analysis Plan (2021-07-21): https://cdn.clinicaltrials.gov/large-docs/60/NCT05016960/SAP_002.pdf